CLINICAL TRIAL: NCT06336018
Title: A Multi-centre, Open-label, Parallel-group Study Investigating the Pharmacokinetics, Safety and Tolerability After a Single Dose of Oral Etavopivat in Participants With Mild, Moderate or Severe Hepatic Impairment Compared to Participants With Normal Hepatic Function
Brief Title: A Research Study on Etavopivat in Participants With and Without Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7535-7703; U1111-1289-2466 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Mild hepatic impairment: Etavopivat dose 2 (Experimental): Participants will receive a single dose of oral etavopivat.
  Interventions: Drug: Etavopivat
- Moderate hepatic impairment: Etavopivat dose 2 (Experimental): Participants will receive a single dose of oral etavopivat.
  Interventions: Drug: Etavopivat
- Healthy matched controls: Etavopivat dose 2 (Experimental): Participants will receive a single dose of oral etavopivat.
  Interventions: Drug: Etavopivat
- Severe hepatic impairment: Etavopivat dose 1 (Experimental): Participants will receive a single dose of oral etavopivat.
  Interventions: Drug: Etavopivat
- Healthy matched controls: Etavopivat dose 1 (Experimental): Participants will receive a single dose of oral etavopivat.
  Interventions: Drug: Etavopivat

INTERVENTIONS:
Drug: Etavopivat — Participants will receive a single dose of etavopivat orally.

SUMMARY:
The study investigates an investigational drug called etavopivat in participants with hepatic impairments and participants with normal hepatic function (matched controls). During the study, all participants will be given a single oral dose of etavopivat. All participants will take the etavopivat orally together with water. After dosing, the study will last for 7 to 9 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age 18 years or above at the time of signing the informed consent.
* Body mass index (BMI) between 18.5 and 42.0 kilogram per meter^2 (kg/m^2) (both inclusive) at screening.
* Body weight greater than or equal to (>=) 40.0 kilogram (kg) at screening.

Specific inclusion criteria only for participants with hepatic impairment:

* Participants with chronic (above 6 months), stable (no significant deterioration in hepatic function in last 2 months as determined by the investigator) hepatic impairment classified as Child-Pugh class A, B or C, as assessed by the investigator and which is confirmed and documented by medical history, physical examination and at least one of the following: hepatic ultrasound, computerised axial tomography (CT) scan, magnetic resonance imaging (MRI), and/or liver biopsy.
* Participants must be on a stable dose of medication and/or treatment regimen (e.g., no expectations of new medications nor changes to current medications within 14 days of dosing).

Specific inclusion criterion only for participants with normal hepatic function:

- Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG), and laboratory safety tests performed during screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive methods.
* Participation (i.e., signed informed consent) in any interventional clinical study within 30 days or 5 times the half-life of the previous investigational medical product (IMP) (if known), whichever is longer, before screening.
* Any disorder, unwillingness or inability, except for conditions associated with hepatic impairment in the group of participants with compromised hepatic function, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Participant is unable to refrain from or anticipates the use of, for 7 days prior to dosing and throughout the study, any drug known to be:

  * an inhibitor of uridine 5'-diphospho-glucuronosyltransferase (UGT) 2B7,
  * a strong inhibitor of cytochrome P450 (CYP)3A4 or CYP2C9,
  * a potent inhibitor of permeability glycoprotein (P-gp).
* Participant is unable to refrain from or anticipates the use of, for 28 days prior to dosing and throughout the study, any drug known to be:

  * an inducer of UGT2B7,
  * a strong or moderate inducer of CYP3A4, including St. John's Wort,
  * a strong inducer of CYP2C9,
  * a potent inducer of P-gp.
* Participant is unable to refrain from or anticipates the use of any medications or substances prohibited in the study.

Specific exclusion criterion only for participants with hepatic impairment:

- Clinical signs of an acute hepatitis (viral as well as non-viral) or positive tests of hepatitis B virus surface antigen (HBsAg) (unless hepatitis B virus titre is negative) or antibody tests of hepatitis C virus (HCV-Ab) (unless negative polymerase chain reaction [PCR] for hepatitis C virus).

Specific exclusion criteria only for participants with normal hepatic function:

* Diagnostic test results positive for hepatitis B or hepatitis C infection.
* History of diabetes mellitus or glycated haemoglobin (HbA1c) greater than or equal to 5 percent (48 millimoles per mole [mmol/mol]) at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Area under the etavopivat plasma concentration-time curve from 0 hours and extrapolated to infinity after a single dose (AUC0-inf, etavopivat) | From IMP administration on day 1 to completion of the end of study visit (day 9)
  Measured in hours*nanogram per milliter (h*ng/mL).
Maximum observed etavopivat plasma concentration after a single dose (Cmax, etavopivat) | From IMP administration on day 1 to completion of the end of study visit (day 9)
  Measured in nanogram per milliter (ng/mL).

SECONDARY OUTCOMES:
Area under the etavopivat plasma concentration-time curve from 0 hours to the last quantifiable concentration after a single dose (AUC0-last, etavopivat) | From IMP administration on day 1 to completion of the end of study visit (day 9)
  Measured in h*ng/mL.
Time to maximum observed etavopivat plasma concentration after a single dose (tmax, etavopivat) | From IMP administration on day 1 to completion of the end of study visit (day 9)
  Measured in hours.
Terminal half-life for etavopivat after a single dose (t1/2, etavopivat) | From IMP administration on day 1 to completion of the end of study visit (day 9)
  Measured in hours.
Apparent plasma clearance of etavopivat after a single dose (CL/Fetavopivat) | From IMP administration on day 1 to completion of the end of study visit (day 9)
  Measured in liter per hour (L/h).
Apparent volume of distribution of etavopivat after a single dose based on plasma concentration values (Vz/Fetavopivat) | From IMP administration on day 1 to completion of the end of study visit (day 9)
  Measured in liter (L).
Number of adverse events (AEs) | From IMP administration on day 1 to completion of the end of study visit (day 9)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Amer. Rrsch Corp-TX Liver Inst, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com